CLINICAL TRIAL: NCT05369442
Title: Prognosis and Antiplatelet Strategies for Patients With PCI and High Bleeding Risk:A Study Protocol
Status: Recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yong He, Professor, cardiology department, principal investigator, West China Hospital
Other Study IDs: WestChinaH-CVD-004
Record Dates: First submitted 2022-04-23; First posted 2022-05-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Percutaneous coronary intervention (PCI) is an important treatment strategy for patients with coronary artery disease. Combined bleeding after PCI significantly increases the risk of death in patients. The search for prognostic predictors and optimal antiplatelet therapy for patients with high bleeding risk (HBR) after PCI has been a hot topic in cardiovascular research. There is no accepted prognostic model or recommended antiplatelet therapy for patients with PCI-HBR. In this project, based on retrospective data extraction and prospective database building, we used artificial intelligence (AI) to analyze the adverse prognostic predictors of PCI-HBR patients, observe the types of antiplatelet drugs and duration of dual antiplatelet therapy in PCI-HBR patients, and compare the safety and feasibility of different antiplatelet regimens and treatment courses. The safety and feasibility of different antiplatelet regimens and regimens were compared.

DETAILED DESCRIPTION:
This trail is a single center investigator-initiated prospective registry. PPP-PCI aims to observe the characteristics and prognosis of the PCI-HBR population and to explore appropriate antiplatelet therapy regimens to provide a basis for intervention guidance for patients with PCI-HBR. This project will help to further improve the existing bleeding prediction models and improve the efficiency of treating PCI-HBR patients.

Patients' baseline information is based on the latest test before PCI procedure. Basic information include age, gender, systolic blood pressure, diastolic blood pressure, body mass index, smoking status, smoking volume, positive family history of cardiovascular disease, hyperlipidemia, hypertension, diabetes, stroke history, peripheral artery disease, etc. Real-time update features include DAPT sessions, MACE event records, symptom records, sign records, test results, diagnosis, medical advice, real-time sign monitoring equipment data, ECG abnormalities, etc. Tests include a full set of lipid levels (including triglycerides, cholesterol, HDL, LDL, etc.), biochemical parameters (including creatinine, glomerular filtration rate, uric acid, etc.), hemoglobin, glucose, glycated hemoglobin, homocysteine, and lipoprotein(a) level. Imaging and functional testing data include coronary angiography images, intervention-related parameters, and target vessel lesion characteristics. The patient data is correlated with the visit intensity. The imaging images are used for deep learning to build unstructured classification models. The non-imaging data are used for machine learning to build a structured classification model. Pre-processing of the data includes image normalization, correction and normalization of irregular values, detection and removal of outliers and anomalies, interpolation and rejection of null values, removal of multicollinearity, and data normalization.

For the imaging images, a deep learning model was constructed using convolutional neural network to dichotomize the coronary vascular lesions and functional conditions contained in the coronary angiography images. For the non-imaging image data, Embedded method was used as the top-level method, and logistic regression, random forest, and gradient boosting tree were used as the bottom-level algorithms, and the key factors affecting the occurrence of MACE in the PCI-HBR population were extracted by fusing the feature weights through integrated learning. Based on the extracted key factors, a binary machine learning discriminative model was established, and SVM, XGBoost, random forest, and artificial neural network were used to complete the evaluation of multiple models, and the best model was selected as the machine learning classification model.

The deep learning model and machine learning model structures are weighted and fused to output the final results. Then the data collected by the future model is passed back to the training dataset for incremental learning to correct the model.

This trial will provide new insights and evidence on optimal antiplatelet therapy for a high bleeding risk patient cohort which is frequently encountered in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

PCI patients >18 years of age and meeting 1 major criterion or 2 minor criteria of the ARC-HBR The ARC-HBR major criteria included:

* long-term use of oral anticoagulants;
* severe or end-stage chronic kidney disease [eGFR <30 ml/(min*1.73m2 )];
* hemoglobin <11 g/dl, spontaneous bleeding requiring hospitalization or transfusion within the past 6 months or at any time;
* chronic bleeding constitutional;
* cirrhosis with portal hypertension spontaneous bleeding requiring hospitalization or transfusion within the past 6 months or at any time;
* moderate to severe baseline thrombocytopenia (platelets <100×10^9/L); chronic bleeding constitutional;
* cirrhosis with portal hypertension;
* active malignancy within the past 12 months (excluding non-melanoma skin cancer);
* previous spontaneous brain hemorrhage (at any time);
* traumatic brain hemorrhage within the past 12 months;
* within the past 6 months moderate or severe ischemic stroke within the past 6 months;
* the presence of cerebral arteriovenous malformation;
* recent major surgery or major trauma within 30 days prior to PCI;
* and major non-delayable surgery during DAPT.

Secondary criteria included:

* age ≥75 years;
* moderate chronic kidney disease [30 ml/(min*1.73m2 ) ≤ eGFR ≤ 59 ml/(min*1.73m2 )];
* 11 g/dl ≤ hemoglobin < 13 g/dl in men and 11 g/dl ≤ hemoglobin < 12 g/dl in women; - spontaneous bleeding requiring hospitalization or blood transfusion in the past 6 months to 12 months;
* long-term use of oral NSAIDs or steroids
* Ischemic stroke of any duration not covered by the primary criteria.

Exclusion Criteria:

* Patients who were already bleeding at the time of baseline inclusion
* Patients who could not be followed up (including previously reserved phone changes, etc.) to obtain MACE events.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: People at high risk of bleeding from PCI who meet one of the primary bleeding risk criteria or two of the secondary bleeding risk criteria, according to the criteria established by the ARC-HBR.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
death | 30 days
  Death will be classified as cardiac or non-cardiac in origin. All causes of death will be considered cardiac unless a clear non-cardiac cause of death can be identified. Of these, hemorrhagic deaths will be specified.
death | 6 months
  Death will be classified as cardiac or non-cardiac in origin. All causes of death will be considered cardiac unless a clear non-cardiac cause of death can be identified. Of these, hemorrhagic deaths will be specified.
death | 1 year
  Death will be classified as cardiac or non-cardiac in origin. All causes of death will be considered cardiac unless a clear non-cardiac cause of death can be identified. Of these, hemorrhagic deaths will be specified.
Myocardial infarction | 30 days
  Defined as recurrent signs or symptoms of myocardial ischemia lasting more than 30 minutes, with new ST-T changes or Q waves in at least two consecutive leads, or new left bundle branch block, and re-elevated cardiac enzyme levels. The following creatine kinase-myocardial band isoenzyme (CK-MB) changes will be considered meaningfully elevated: CK-MB elevation on the basis of a ≥25% decrease in peak; CK-MB elevation >50% from the previous elevation; CK-MB elevation >2 times the normal upper limit in non-coronary interventions; CK-MB elevation >2 times the normal upper limit after PCI. CK-MB is greater than 5 times the upper limit of normal after PCI.
Myocardial infarction | 6 months
  Defined as recurrent signs or symptoms of myocardial ischemia lasting more than 30 minutes, with new ST-T changes or Q waves in at least two consecutive leads, or new left bundle branch block, and re-elevated cardiac enzyme levels. The following creatine kinase-myocardial band isoenzyme (CK-MB) changes will be considered meaningfully elevated: CK-MB elevation on the basis of a ≥25% decrease in peak; CK-MB elevation >50% from the previous elevation; CK-MB elevation >2 times the normal upper limit in non-coronary interventions; CK-MB elevation >2 times the normal upper limit after PCI. CK-MB is greater than 5 times the upper limit of normal after PCI.
Myocardial infarction | 1 year
  Defined as recurrent signs or symptoms of myocardial ischemia lasting more than 30 minutes, with new ST-T changes or Q waves in at least two consecutive leads, or new left bundle branch block, and re-elevated cardiac enzyme levels. The following creatine kinase-myocardial band isoenzyme (CK-MB) changes will be considered meaningfully elevated: CK-MB elevation on the basis of a ≥25% decrease in peak; CK-MB elevation >50% from the previous elevation; CK-MB elevation >2 times the normal upper limit in non-coronary interventions; CK-MB elevation >2 times the normal upper limit after PCI. CK-MB is greater than 5 times the upper limit of normal after PCI.
Ischemic stroke | 30 days, 6 months, 1 year
  Acute onset of focal or global neurological deficits lasting more than 24 hours, confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) as ischemic stroke
Ischemic stroke | 30 days
  Acute onset of focal or global neurological deficits lasting more than 24 hours, confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) as ischemic stroke
Ischemic stroke | months
  Acute onset of focal or global neurological deficits lasting more than 24 hours, confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) as ischemic stroke
Ischemic stroke | 1 year
  Acute onset of focal or global neurological deficits lasting more than 24 hours, confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) as ischemic stroke
Major bleeding | 30 days, 6 months, 1 year
  The severity of bleeding is graded according to the BARC criteria recommended by the International Society for the Study of Hemorrhage, and the site of bleeding is described, including intracranial, gastrointestinal, respiratory (e.g., hemoptysis), urinary (e.g., hematuria), subcutaneous or mucosal, gingival, nasal, ophthalmic, and surgical puncture site related. Minor bleeds are BARC types 1 and 2, and major bleeds are BARC types 3 and 5.
Major bleeding | 30 days
  The severity of bleeding is graded according to the BARC criteria recommended by the International Society for the Study of Hemorrhage, and the site of bleeding is described, including intracranial, gastrointestinal, respiratory (e.g., hemoptysis), urinary (e.g., hematuria), subcutaneous or mucosal, gingival, nasal, ophthalmic, and surgical puncture site related. Minor bleeds are BARC types 1 and 2, and major bleeds are BARC types 3 and 5.
Major bleeding | 6 months
  The severity of bleeding is graded according to the BARC criteria recommended by the International Society for the Study of Hemorrhage, and the site of bleeding is described, including intracranial, gastrointestinal, respiratory (e.g., hemoptysis), urinary (e.g., hematuria), subcutaneous or mucosal, gingival, nasal, ophthalmic, and surgical puncture site related. Minor bleeds are BARC types 1 and 2, and major bleeds are BARC types 3 and 5.
Major bleeding | 1 year
  The severity of bleeding is graded according to the BARC criteria recommended by the International Society for the Study of Hemorrhage, and the site of bleeding is described, including intracranial, gastrointestinal, respiratory (e.g., hemoptysis), urinary (e.g., hematuria), subcutaneous or mucosal, gingival, nasal, ophthalmic, and surgical puncture site related. Minor bleeds are BARC types 1 and 2, and major bleeds are BARC types 3 and 5.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Sichuan, Sichuan, China

REFERENCES:
- [Derived] Zhang J, Chen Z, Liu R, Li Y, Zhao H, Li Y, Zhou M, Wang H, Li C, Rao L, He Y. Development and Validation of a Nomogram for Predicting Long-Term Net Adverse Clinical Events in High Bleeding Risk Patients Undergoing Percutaneous Coronary Intervention. Rev Cardiovasc Med. 2025 Jan 17;26(1):25352. doi: 10.31083/RCM25352. eCollection 2025 Jan. PMID 39867174